CLINICAL TRIAL: NCT07112066
Title: Natural History of Cardiac Transthyretin Amyloidosis - Mechanistic Insights by Multimodality Imaging
Brief Title: Multimodality Cardiac Imaging for Disease Progression in ATTR-CM
Acronym: FAPI-ATTR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dominik Benz (Other)
Collaborators: Olga Mayenfisch Stiftung, Zurich, Switzerland (Unknown); University of Zurich (Other)
Responsible Party: Sponsor-Investigator, Dominik Benz, PD Dr. med. Dominik C. Benz, University of Zurich
Organization: University of Zurich (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2024-02504
Record Dates: First submitted 2025-07-14; First posted 2025-08-08 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Amyloidosis Cardiac
Keywords: cardiac ATTR amyloidosis; BMP4 protein, human; 18F-FAPI-74; PET; CT
MeSH Terms: conditions — Amyloid Neuropathies, Familial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 18F-FAPI PET/CT (Experimental): Additional imaging including 18F-FAPI PET/CT is performed
  Interventions: Diagnostic Test: FAPI tracer

INTERVENTIONS:
Diagnostic Test: FAPI tracer — 18F-FAPI-74 PET/CT, cardiac MRI, echocardiography and blood sample for BMP5 serum concetration is performed at baseline and 12-month follow-up.

SUMMARY:
The goal of this clinical trial is to investigate whether new imaging techniques can help us to better understand the cardiac amyloidosis. The disease can be slowed down with various medications (e.g., tafamidis, acoramidis, or vutrisiran). However, treatment is not effective in all patients-in about one-third of cases, the disease continues to progress. So far, we know little about the exact causes of this and what biological changes occur in the heart muscle.

The main question it aims to answer is:

Will new imaging techniques help us understand the course of the cardiac amyloidosis?

Participants will have additional examinations:

* At the beginning of the study: one additional heart ultrasound examination, one cardiac MRI and one cardiac PET, blood examination during the regular examination, questionnaires.
* After a year: one additional heart ultrasound examination, one cardiac MRI and one cardiac PET, blood examination during the regular examination.

Time required:

* Heart ultrasound examination: 5-10 Minutes
* Cardiac MRI: 2 hours
* Cardiac PET: 2 hours
* Questionnaires: 5-10 Minutes.

DETAILED DESCRIPTION:
Experimental Design The study design is an open label prospective longitudinal study with serial imaging at baseline and after 12-month follow-up. The entire study population will include 50 participants with cardiac ATTR amyloidosis, as recently defined by multi-societal criteria.

Conventional markers of disease progression

These markers are collected during routine clinical follow-up of patients in our Outpatient Clinic. The markers are divided into three domains and include the following outcomes:

* Clinical and functional: any heart failure hospitalization, NYHA class, Kansas City Cardiomyopathy Questionnaire, 6-minute walk test;
* Laboratory biomarkers: NT-proBNP, troponin, creatinine;
* Imaging and ECG: LV wall thickness, diastolic dysfunction, LVEF, stroke volume, global longitudinal strain, conduction disturbance.

Data Analysis Plan Power calculation for sample size is challenging as no previous study has evaluated the response of our endpoints in myocardial FAPI uptake or serum BMP4 concentration to tafamidis. We therefore focused sample size calculation of echocardiographic myocardial stiffness. Based on our own preliminary data, we estimate median baseline values for myocardial stiffness of 2.6 m/s [IQR, 1.7-3.8] in cardiac amyloidosis. Disease progression is expected in about 30% of participants. While myocardial stiffness is expected to remain unchanged in cardiac amyloidosis without disease progression a 20% relative increase (i.e. 0.5 ± 0.5 m/s) is considered in cardiac amyloidosis with disease progression. A sample size of 40 participants (i.e. 30 participants without and 10 participants with disease progression) has a statistical power of 80% to predict a difference in response of myocardial stiffness to tafamidis.

Non-normally distributed, paired data of repeated measures (i.e. longitudinal changes per group) are compared by Wilcoxon signed rank test. Non-normally distributed unpaired data of changes (i.e. longitudinal changes between groups) are compared by Mann-Whitney test. The correlations are compared by a z-test on Fisher z-transformed correlation coefficients.

ELIGIBILITY:
Inclusion Criteria:

* Participants with cardiac ATTR amyloidosis, as recently defined by multi-societal criteria, who are about to start tafamidis at the University Hospital Zurich

Exclusion Criteria:

* Any other disease-modifying therapy (e.g. patisiran)
* Ongoing supraventricular arrhythmia
* Ventricular pacing
* Prior septal myocardial infarction

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-10-20 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Change in FAPI uptake | Baseline and 1 year
  F-FAPI-74 PET/CT is performed at baseline and 12-month follow-up. Images are acquired on a PET/CT scanner 60 minutes after intravenous injection of F-FAPI-74. The emission scan is obtained from the apex of the lung to the base of the lung. One bed position is acquired (20 minutes, 3-dimensional mode), and the heart is set at the center of the view. Myocardial F-FAPI-74 uptake is quantified by the mean standardized uptakte value of the LV volume of interest (VOI). The epicardial LV contour is drawn on the CT scan and, to correct for blood pool activity, the endocardial border is defined automatically by thresholding for 2 times the mean SUV of the blood pool.

SECONDARY OUTCOMES:
Change in echocardiographic myocardial stiffness | Baseline and 1 year
  Cardiac intrinsic elastography from echocardiography is performed at baseline and at 12-month follow-up. Ultrahigh-frame rate tissue Doppler data (>250 frames/sec) are acquired using clinical scanners from the apical fourchamber view while carefully aligning the septal wall with the Doppler beam. The base-to-apex propagation of the late diastolic myocardial stretch wave can be visualized with ultrafast imaging data. The slope of the isovelocity wave front, called intrinsic velocity propagation (iVP) of myocardial stretch (in meters per second) is measured offline. By averaging values for three cardiac cycles, a global value is generated.
Change in extracellular volume (ECV) | Baseline and 1 year
  Cardiac MRI is performed at baseline and 12-month follow-up. Myocardial LV native T1 maps are acquired in 3 short-axis slices at the base, mid and apical levels using the modified Look-Locker inversion (MOLLI) recovery technique at end-diastole for 3 cycles (5-3-1 R-R durations with 3-4 R-R rest periods) during a single breath hold. T1 mapping is repeated with the same settings 10 minutes after intravenous administration of 0.1 mmol/kg of gadolinium contrast agent. The ECV fraction is estimated by plotting the reciprocal of each segmental myocardial T1 against the reciprocal of the blood pool T1 for native, 10-minute post-contrast MOLLI acquisitions, then calculating linear regression slopes, corresponding to segmental partition coefficients for gadolinium (λGd). Each λGd was multiplied by (1 - hematocrit) to obtain ECV fractions.
Change in BMP4 expression and serum concentration | Baseline and 1 year
  Serum samples are analyzed. BMP4 levels in the samples were measured using a human BMP4 SimpleStep ELISA Kit following manufacturer's instructions.
  Endomyocardial biopsies as part of the clinical diagnostic routine from the subgroup of 10 participants with suspicion of cardiac ATTR amyloidosis are analyzed. Cardiac tissue is fixed in 4% formaladehyde and embedded in paraffin. Histopathological changes are evaluated after H&E staining and the area of percentage of collagen networks per section is determined. For the assessment of BMP4 mRNA expression in tissue, homogenates are generated, samples are centrifuged and the supernatant is used for ELISA measurements.

CONTACTS AND LOCATIONS:
Overall Officials: Dominik C Benz, MD, Principal Investigator — Universität Zürich
Locations (1):
- University Hospital Zurich, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No